CLINICAL TRIAL: NCT05762302
Title: A Multicenter Randomized Controlled Trial to Establish the Impact of MeMed BV® on Management of Patients With Suspected Lower Respiratory Tract Infections (LRTI) in the Emergency Department (ED) and Urgent Care Center (UCC) ("JUPITER" TRIAL)
Brief Title: The Impact of MeMed BV® on Management of Patients With Suspected Lower Respiratory Tract Infections (LRTI) in the Emergency Department (ED) and Urgent Care Center (UCC) ("JUPITER" TRIAL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MMD013RCT
Record Dates: First submitted 2023-02-13; First posted 2023-03-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lower Respiratory Tract Infection

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: applicable only for control arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Adults with suspected Lower Respiratory Track Infection (LRTI)- The MeMed BV arm (Experimental): ED and urgent care center patients over the age of 18 years , with clinical suspicion of Lower Respiratory Track Infection. clinician will receive the BV result, this will include a recommendation regarding antibiotic treatment. A telephone FU call will be done at 28 (+/- 3) days after the day of consent to complete a short questionnaire regarding your current illness
  Interventions: Diagnostic Test: MeMed BV test
- Adults with suspected Lower Respiratory Track Infection (LRTI)- The control arm (No Intervention): ED and urgent care center patients over the age of 18 years , with clinical suspicion of Lower Respiratory Track Infection. clinician will not receive the BV result, and will treat according to standard of care. A telephone FU call will be done at 28 (+/- 3) days after the day of consent to complete a short questionnaire regarding your current illness

INTERVENTIONS:
Diagnostic Test: MeMed BV test — Following the MeMed BV test result, the clinician will decide whether or not to prescribe an antibiotic for your condition
  Arms: Adults with suspected Lower Respiratory Track Infection (LRTI)- The MeMed BV arm

SUMMARY:
This is a Prospective, multi-center study enrolling adults subjects presented to the ED/Urgent care, with symptoms consistent with lower respiratory infection (LRTI).

The reason of this study is to demonstrate the MeMed BV can help clinicians make decisions about using antibiotics in patients with lower respiratory track infections and see how it would impact clinical outcomes, antibiotics use, hospitalizations, ED clinicians find ways to improve health and medical care.

DETAILED DESCRIPTION:
There will be a pre-study implementation phase (JUNO trial), in which approximately 250 patients will be recruited. Data obtained for these patients will not be included in the analysis. The purpose of the pre-study implementation phase is to enable the participating clinicians to become familiar with the MeMed BV test. An additional purpose is to test the design and operational assumptions before the subsequent JUPITER trial.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients eligible for inclusion are required to fulfill all of the following criteria:
* Written informed consent must be obtained from the patient or his/her legal guardian.
* 18 years of age or older.
* Current disease duration ≤ 7 days.
* Tactile fever or measured temperature ≥ 37.8°C (100°F) (any body site, any measurement device, including self-reported), either of them noted at least once within the last 7 days.
* Clinical suspicion of bacterial or viral LRTI: At least one of the following respiratory signs or symptoms: cough (new or worsening), sputum production, dyspnea/shortness of breath, auscultatory abnormality (e.g. wheezing, rhonchi).
* Clinician intent to prescribe antibiotics based on the currently available data.

EXCLUSION CRITERIA

Patients fulfilling any of the following criteria are not eligible for inclusion in the infectious cohort:

* Systemic antibiotics within 72 hours prior to enrollment
* Inflammatory disease (e.g., IBD, SLE, Rheumatoid arthritis, Kawasaki, other vasculitis)
* Congenital immune deficiency (CID)
* A proven or suspected infection on presentation with Mycobacterial (e.g., MAC, MABC), parasitic or fungal (e.g., Candida, Histoplasma, Aspergillus) pathogen
* HIV, HBV, or HCV infection (self-declared or known from medical records)
* Major surgery, trauma and\or burns in the last 7 days
* Pregnancy- self reported or medically confirmed
* Active malignancy - Cancer diagnosed within the previous six months, recurrent, regionally advanced or metastatic cancer, cancer for which treatment had been administered within six months, or hematological cancer that is not in complete remission.
* Patients with severe illnesses that affect life expectancy and quality of life such as end stage renal disease, end stage liver disease or severe COPD.
* Clinician intent to hospitalize patient.
* Patients with suspected concomitant infections (e.g. UTI, cellulitis, gastroenteritis, etc.)
* Active treatment with immune-suppressive or immune-modulating therapies, including without limitations:

Administration of PO\IV\IM high dose steroids >1mg/kg/day prednisone (or equivalent) at some point in the past 10 days or daily continuous use of steroids > 0.25 mg/kg/day in the past 7 days Monoclonal antibodies, anti-TNF agents Intravenous immunoglobulin (IVIG) Cyclosporine, Cyclophosphamide, Tacrolimus, Azathioprine, Methotrexate G/GM-CSF, Interferons

•Considered unsuitable for the study by the study team

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1316 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
To demonstrate MeMed BV® added value on top of standard of care in lowering unwarranted antibiotic prescribing in patients with LRTI in the ED/UCC. | Through study completion, an average of 18 months
  Primary outcome is total antibiotic prescription in the ED/UCC in the BV and control arms, defined as antibiotic initiation by the initial ED/UCC clinician (reached if the patient received antibiotics during ED/UCC visit).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - University of Florida-Jacksonville, Jacksonville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Maimonides Medical Center, Brooklyn, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Philadelphia Thomas Jefferson ED, Philadelphia, Pennsylvania
  - Medical University South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - MCW, Milwaukee, Wisconsin
- Israel (2):
  - Carmel Medical Center, Haifa, North
  - Lin Medical Center, Haifa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Antimicrobial Resistance Collaborators. Global burden of bacterial antimicrobial resistance in 2019: a systematic analysis. Lancet. 2022 Feb 12;399(10325):629-655. doi: 10.1016/S0140-6736(21)02724-0. Epub 2022 Jan 19. PMID 35065702
- [Result] Prestinaci F, Pezzotti P, Pantosti A. Antimicrobial resistance: a global multifaceted phenomenon. Pathog Glob Health. 2015;109(7):309-18. doi: 10.1179/2047773215Y.0000000030. Epub 2015 Sep 7. PMID 26343252
- [Result] Jourdan A, Sangha B, Kim E, Nawaz S, Malik V, Vij R, Sekhsaria S. Antibiotic hypersensitivity and adverse reactions: management and implications in clinical practice. Allergy Asthma Clin Immunol. 2020 Jan 21;16:6. doi: 10.1186/s13223-020-0402-x. eCollection 2020. PMID 31993070
- [Result] Lovegrove MC, Geller AI, Fleming-Dutra KE, Shehab N, Sapiano MRP, Budnitz DS. US Emergency Department Visits for Adverse Drug Events From Antibiotics in Children, 2011-2015. J Pediatric Infect Dis Soc. 2019 Nov 6;8(5):384-391. doi: 10.1093/jpids/piy066. PMID 30137509
- [Result] Tamma PD, Avdic E, Li DX, Dzintars K, Cosgrove SE. Association of Adverse Events With Antibiotic Use in Hospitalized Patients. JAMA Intern Med. 2017 Sep 1;177(9):1308-1315. doi: 10.1001/jamainternmed.2017.1938. PMID 28604925
- [Result] Nelson RE, Hatfield KM, Wolford H, Samore MH, Scott RD, Reddy SC, Olubajo B, Paul P, Jernigan JA, Baggs J. National Estimates of Healthcare Costs Associated With Multidrug-Resistant Bacterial Infections Among Hospitalized Patients in the United States. Clin Infect Dis. 2021 Jan 29;72(Suppl 1):S17-S26. doi: 10.1093/cid/ciaa1581. PMID 33512523
- [Result] Cassini A, Hogberg LD, Plachouras D, Quattrocchi A, Hoxha A, Simonsen GS, Colomb-Cotinat M, Kretzschmar ME, Devleesschauwer B, Cecchini M, Ouakrim DA, Oliveira TC, Struelens MJ, Suetens C, Monnet DL; Burden of AMR Collaborative Group. Attributable deaths and disability-adjusted life-years caused by infections with antibiotic-resistant bacteria in the EU and the European Economic Area in 2015: a population-level modelling analysis. Lancet Infect Dis. 2019 Jan;19(1):56-66. doi: 10.1016/S1473-3099(18)30605-4. Epub 2018 Nov 5. PMID 30409683
- [Result] Fendrick AM, Monto AS, Nightengale B, Sarnes M. The economic burden of non-influenza-related viral respiratory tract infection in the United States. Arch Intern Med. 2003 Feb 24;163(4):487-94. doi: 10.1001/archinte.163.4.487. PMID 12588210
- [Result] Bartlett JG. Clinical practice. Antibiotic-associated diarrhea. N Engl J Med. 2002 Jan 31;346(5):334-9. doi: 10.1056/NEJMcp011603. No abstract available. PMID 11821511
- [Result] Giannelli FR. Antibiotic-associated diarrhea. JAAPA. 2017 Oct;30(10):46-47. doi: 10.1097/01.JAA.0000524721.01579.c9. No abstract available. PMID 28953024
- [Result] Collins AM, Johnstone CM, Gritzfeld JF, Banyard A, Hancock CA, Wright AD, Macfarlane L, Ferreira DM, Gordon SB. Pneumococcal Colonization Rates in Patients Admitted to a United Kingdom Hospital with Lower Respiratory Tract Infection: a Prospective Case-Control Study. J Clin Microbiol. 2016 Apr;54(4):944-9. doi: 10.1128/JCM.02008-15. Epub 2016 Jan 20. PMID 26791364
- [Result] Lim YK, Kweon OJ, Kim HR, Kim TH, Lee MK. Impact of bacterial and viral coinfection in community-acquired pneumonia in adults. Diagn Microbiol Infect Dis. 2019 May;94(1):50-54. doi: 10.1016/j.diagmicrobio.2018.11.014. Epub 2018 Nov 24. PMID 30578007
- [Result] Rao S, Lamb MM, Moss A, Mistry RD, Grice K, Ahmed W, Santos-Cantu D, Kitchen E, Patel C, Ferrari I, Dominguez SR. Effect of Rapid Respiratory Virus Testing on Antibiotic Prescribing Among Children Presenting to the Emergency Department With Acute Respiratory Illness: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jun 1;4(6):e2111836. doi: 10.1001/jamanetworkopen.2021.11836. PMID 34086034
- [Result] Herberg JA, Kaforou M, Gormley S, Sumner ER, Patel S, Jones KD, Paulus S, Fink C, Martinon-Torres F, Montana G, Wright VJ, Levin M. Transcriptomic profiling in childhood H1N1/09 influenza reveals reduced expression of protein synthesis genes. J Infect Dis. 2013 Nov 15;208(10):1664-8. doi: 10.1093/infdis/jit348. Epub 2013 Jul 29. PMID 23901082
- [Result] Wong JG, Aung AH, Lian W, Lye DC, Ooi CK, Chow A. Risk prediction models to guide antibiotic prescribing: a study on adult patients with uncomplicated upper respiratory tract infections in an emergency department. Antimicrob Resist Infect Control. 2020 Nov 2;9(1):171. doi: 10.1186/s13756-020-00825-3. PMID 33138859
- [Result] de la Poza Abad M, Mas Dalmau G, Moreno Bakedano M, Gonzalez Gonzalez AI, Canellas Criado Y, Hernandez Anadon S, Rotaeche del Campo R, Toran Monserrat P, Negrete Palma A, Munoz Ortiz L, Borrell Thio E, Llor C, Little P, Alonso-Coello P; Delayed Antibiotic Prescription (DAP) Group. Prescription Strategies in Acute Uncomplicated Respiratory Infections: A Randomized Clinical Trial. JAMA Intern Med. 2016 Jan;176(1):21-9. doi: 10.1001/jamainternmed.2015.7088. PMID 26719947
- [Result] Rowe TA, Linder JA. Novel approaches to decrease inappropriate ambulatory antibiotic use. Expert Rev Anti Infect Ther. 2019 Jul;17(7):511-521. doi: 10.1080/14787210.2019.1635455. Epub 2019 Jul 5. PMID 31232615
- [Result] Huang DT, Yealy DM, Filbin MR, Brown AM, Chang CH, Doi Y, Donnino MW, Fine J, Fine MJ, Fischer MA, Holst JM, Hou PC, Kellum JA, Khan F, Kurz MC, Lotfipour S, LoVecchio F, Peck-Palmer OM, Pike F, Prunty H, Sherwin RL, Southerland L, Terndrup T, Weissfeld LA, Yabes J, Angus DC; ProACT Investigators. Procalcitonin-Guided Use of Antibiotics for Lower Respiratory Tract Infection. N Engl J Med. 2018 Jul 19;379(3):236-249. doi: 10.1056/NEJMoa1802670. Epub 2018 May 20. PMID 29781385
- [Result] Oved K, Cohen A, Boico O, Navon R, Friedman T, Etshtein L, Kriger O, Bamberger E, Fonar Y, Yacobov R, Wolchinsky R, Denkberg G, Dotan Y, Hochberg A, Reiter Y, Grupper M, Srugo I, Feigin P, Gorfine M, Chistyakov I, Dagan R, Klein A, Potasman I, Eden E. A novel host-proteome signature for distinguishing between acute bacterial and viral infections. PLoS One. 2015 Mar 18;10(3):e0120012. doi: 10.1371/journal.pone.0120012. eCollection 2015. PMID 25785720
- [Result] Herberg JA, Kaforou M, Wright VJ, Shailes H, Eleftherohorinou H, Hoggart CJ, Cebey-Lopez M, Carter MJ, Janes VA, Gormley S, Shimizu C, Tremoulet AH, Barendregt AM, Salas A, Kanegaye J, Pollard AJ, Faust SN, Patel S, Kuijpers T, Martinon-Torres F, Burns JC, Coin LJ, Levin M; IRIS Consortium. Diagnostic Test Accuracy of a 2-Transcript Host RNA Signature for Discriminating Bacterial vs Viral Infection in Febrile Children. JAMA. 2016 Aug 23-30;316(8):835-45. doi: 10.1001/jama.2016.11236. PMID 27552617
- [Result] Lydon EC, Henao R, Burke TW, Aydin M, Nicholson BP, Glickman SW, Fowler VG, Quackenbush EB, Cairns CB, Kingsmore SF, Jaehne AK, Rivers EP, Langley RJ, Petzold E, Ko ER, McClain MT, Ginsburg GS, Woods CW, Tsalik EL. Validation of a host response test to distinguish bacterial and viral respiratory infection. EBioMedicine. 2019 Oct;48:453-461. doi: 10.1016/j.ebiom.2019.09.040. Epub 2019 Oct 17. PMID 31631046
- [Result] Srugo I, Klein A, Stein M, Golan-Shany O, Kerem N, Chistyakov I, Genizi J, Glazer O, Yaniv L, German A, Miron D, Shachor-Meyouhas Y, Bamberger E, Oved K, Gottlieb TM, Navon R, Paz M, Etshtein L, Boico O, Kronenfeld G, Eden E, Cohen R, Chappuy H, Angoulvant F, Lacroix L, Gervaix A. Validation of a Novel Assay to Distinguish Bacterial and Viral Infections. Pediatrics. 2017 Oct;140(4):e20163453. doi: 10.1542/peds.2016-3453. Epub 2017 Sep 13. PMID 28904072
- [Result] van Houten CB, de Groot JAH, Klein A, Srugo I, Chistyakov I, de Waal W, Meijssen CB, Avis W, Wolfs TFW, Shachor-Meyouhas Y, Stein M, Sanders EAM, Bont LJ. A host-protein based assay to differentiate between bacterial and viral infections in preschool children (OPPORTUNITY): a double-blind, multicentre, validation study. Lancet Infect Dis. 2017 Apr;17(4):431-440. doi: 10.1016/S1473-3099(16)30519-9. Epub 2016 Dec 22. PMID 28012942
- [Result] Papan C, Argentiero A, Porwoll M, Hakim U, Farinelli E, Testa I, Pasticci MB, Mezzetti D, Perruccio K, Etshtein L, Mastboim N, Moscoviz E, Ber TI, Cohen A, Simon E, Boico O, Shani L, Gottlieb TM, Navon R, Barash E, Oved K, Eden E, Simon A, Liese JG, Knuf M, Stein M, Yacobov R, Bamberger E, Schneider S, Esposito S, Tenenbaum T. A host signature based on TRAIL, IP-10, and CRP for reducing antibiotic overuse in children by differentiating bacterial from viral infections: a prospective, multicentre cohort study. Clin Microbiol Infect. 2022 May;28(5):723-730. doi: 10.1016/j.cmi.2021.10.019. Epub 2021 Nov 10. PMID 34768022
- [Derived] Singer AJ, Hollander JE, Kean ER, Ring H, Peacock WF, Soto-Ruiz KM, Motov S, Thoppil J, Hendry P, Halabi S, Meltzer AC, Headden GF, Brosh-Nissimov T, Zeltser D, Cannon CM. Effect of host-protein test (TRAIL/IP-10/CRP) on antibiotic prescription and emergency department or urgent care center return visits: The JUNO pilot randomized controlled trial. Acad Emerg Med. 2025 Sep;32(9):975-984. doi: 10.1111/acem.70031. Epub 2025 Apr 18. PMID 40251855
- See also: Antimicrobial resistance — https://www.who.int/news-room/fact-sheets/detail/antimicrobial-resistance
- See also: Tackling drug-resistant infections globally: final report and recommendations — https://amr-review.org/sites/default/files/160518_Final%20paper_with%20cover.pdf
- See also: A generalizable 29-mRNA neural-network classifier for acute bacterial and viral infections — https://www.nature.com/articles/s41467-020-14975-w